CLINICAL TRIAL: NCT04041089
Title: Development and Evaluation of the Effectiveness of Rehabilitation Tools for Neurovisual Disorders in Patients With Posterior Cortical Atrophy (PCA)
Brief Title: Development of the Effectiveness of Rehabilitation Tools for Neurovisual Disorders in Patients With Posterior Cortical Atrophy
Acronym: REEDUC-ACP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-AOI-02
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-02

CONDITIONS: Posterior Cortical Atrophy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Recognition of objects (Experimental): Patients will do the therapy in the following order: object location, object manipulation and object recognition
  Interventions: Behavioral: Recognition of objects
- Location of objects (Experimental): Patients will do the therapy in the following order: object recognition, object location, and object manipulation
  Interventions: Behavioral: Location of objects
- Manipulation of objects (Experimental): Patients will do the therapy in the following order: object manipulation, object recognition and object location
  Interventions: Behavioral: Manipulation of objects

INTERVENTIONS:
Behavioral: Recognition of objects — * Name of shapes / colors / images / objects
  * Classification of shapes / colors / images / objects
  Arms: Recognition of objects
Behavioral: Location of objects — * Search for frequent/rarse targets among distractors sharing one or more characteristics with the target
  * Hit/catch a stationary/mobile target as quickly as possible
  Arms: Location of objects
Behavioral: Manipulation of objects — * Storage of shapes/objects
  * Use of everyday objects (pen, cutlery, etc.)
  Arms: Manipulation of objects

SUMMARY:
Posterior cortical atrophy (PCA) is manifested by neuro-visual disorders that alter the spatial location of objects, their manipulation and/or recognition. Its etiology is most often neurodegenerative, with a major impact on the autonomy and mood of patients and their families. Few studies have focused on non-medication management of these disorders.

The present study thus has a double objective: the development of a complete tool to work on the recognition, localization and/or manipulation of objects; and the evaluation of the effectiveness of this type of management.

ELIGIBILITY:
Inclusion Criteria:

* Age >50 years old
* Male or Female
* Patients with a diagnosis of PCA according to the criteria of Tang-Wai et al (2004)
* MMS>15
* Voluntary, written and informed consent of the patient himself or its legal representative (guardian/curator), with oral consent of the patient in all cases
* Anti-Alzheimer's and psychotropic treatments stable for one month, if taken by the patient
* Affiliation to a social security system

Exclusion Criteria:

* Uncorrected visual disorders with non-degenerative etiology (AV<0.5)
* Person under the protection of justice
* Pregnant women (a pregnancy test will be performed in premenopausal women)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Effectiveness evaluation | At week 34
  Effectiveness will be evaluated a score based on success rate (from 0 to 10), reaction time and eye-recording .

CONTACTS AND LOCATIONS:
Overall Officials: MOUTON Aurélie, Ph, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Institut Claude Pompidou - Centre Mémoire de Ressources et de Recherche du CHU de Nice, Nice, Alpes-Maritime, France

IPD SHARING:
Plan to Share IPD: No